CLINICAL TRIAL: NCT00562406
Title: Ranibizumab for Branch Retinal Vein Occlusion Associated Macular Edema Study (RABAMES)
Acronym: RABAMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinikum Ludwigshafen (Other)
Collaborators: Norvartis Pharma, Nuremberg, Germany (Unknown); Coordination center for clinical studies, Mainz, Germany (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-06104G
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Macular Edema
Keywords: Macular edema secondary to branch retinal vein occlusion
MeSH Terms: conditions — Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): laser photocoagulation to the retina at the area of edema
  Interventions: Procedure: Laser photocoagulation
- 2 (Experimental): intravitreal injection of ranibizumab
  Interventions: Drug: Ranibizumab; Procedure: Laser photocoagulation
- 3 (Experimental): laser photocoagulation to the retina at the area of edema and intravitreal injection of ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — intravitreal injection of 0.5 mg ranibizumab after randomisation, at week 4 and 8
  Other Names: Lucentis
  Arms: 2; 3
Procedure: Laser photocoagulation — laser photocoagulation to the retina at the area of edema
  Arms: 1; 2

SUMMARY:
The primary objective of this pilot study is to compare the functional and anatomic outcomes of chronic macular edema secondary to branch retinal vein occlusion (BRVO) treated with argon laser photocoagulation versus intravitreal ranibizumab (Lucentis®) injection versus a combination of both.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older with chronic (> 3months, < 18 months) macular edema secondary to branch retinal vein occlusion
* Patients who at baseline have a BSCVA in the study eye between 20/320 and equivalent to 20/40, using an ETDRS chart measured at 4 meters
* Patients who at baseline have a chronic macular edema (> 3 months) in the study eye with the following characteristics as determined by fluorescein angiography:
* Evidence that the macular edema extends under the geometric center of the foveal avascular zone.
* Evidence that the edema is only secondary to BRVO (no other relevant ocular diseases, e.g. uveitis).
* Patients who at baseline have a chronic macular edema (> 3 months) in the study eye with the following characteristics as determined by optical coherence tomography (OCT 3):
* Evidence that central macular thickness is > 225 μm.
* Ability of subject to understand character and individual consequences of clinical trial.
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures.
* For women with childbearing potential, adequate contraception (negative pregnancy test result, serum or urine at trial entry, after treatment and at end of study).
* Only one eye of a patient may be included to this trial.

Exclusion Criteria:

* Patients who at baseline
* Have a relevant ocular disease which may be associated with increased intraocular VEGF levels (namely uveitis, neovascular glaucoma, neovascular age-related macular degeneration, diabetic retinopathy, diabetic maculopathy, ocular ischemic syndrome, and others)
* Have a relevant systemic disease which may be associated with increased systemic VEGF levels (namely all malignancies)
* Had previous treatment for macular edema (laser, triamcinolone, vitrectomy)
* Pregnancy and lactation.
* History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
* Participation in other clinical trials within the last 3 months.
* Medical or psychological condition that would not permit completion of the trial or signing of informed consent.
* Arterial hypertension refractory to medical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in best spectacle-corrected visual acuity (BSCVA) | from baseline to month 6

SECONDARY OUTCOMES:
Mean change in BSCVA | from baseline to month 3
Proportion of patients who gain ≥ 5, 10, 15 letters of BSCVA | from baseline to month 3 and 6
Proportion of patients who lose less than 15 letters of BCVA | from baseline to month 3 and 6
Change in area and intensity of leakage | from baseline to month 1, 3 and 6
Mean change in central macular thickness (by OCT) | from baseline to month 1, 3 and 6
Mean change in central macular thickness (by OCT) | from month 3 to 6

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olof Hattenbach, MD, Privatdozent, Principal Investigator — Dept. of Ophthalmology, Ludwigshafen hospital
Locations (4):
- Germany (4):
  - RABAMES investigational trial site, Freiburg im Breisgau
  - RABAMES investigational trial site, Göttingen
  - RABAMES investigational trial site, Ludwigshafen
  - RABAMES investigational trial site, Mainz

REFERENCES:
- [Derived] Pielen A, Mirshahi A, Feltgen N, Lorenz K, Korb C, Junker B, Schaefer C, Zwiener I, Hattenbach LO; RABAMES Study Group. Ranibizumab for Branch Retinal Vein Occlusion Associated Macular Edema Study (RABAMES): six-month results of a prospective randomized clinical trial. Acta Ophthalmol. 2015 Feb;93(1):e29-37. doi: 10.1111/aos.12488. Epub 2014 Jul 8. PMID 25042729